CLINICAL TRIAL: NCT02675868
Title: The Effects of Different Vasopressors on the Innate Immune Response During Experimental Human Endotoxemia, a Pilot Proof-of-principle Study
Brief Title: Effects of Vasopressors on Immune Response
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NL53411.091.015
Record Dates: First submitted 2016-01-25; First posted 2016-02-05 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-04

CONDITIONS: Endotoxemia
Keywords: noradrenaline; vasopressin; phenylephrine; endotoxemia; Lipopolysaccharide; vasopressor
MeSH Terms: conditions — Endotoxemia; Diabetes Insipidus | interventions — Norepinephrine; Phenylephrine; Vasopressins; Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Norepinephrine (Experimental): The noradrenaline group: a group of 10 subjects that will receive noradrenaline 0.05 μg/kg/min infusion for 5 hours, starting 60 minutes before endotoxin administration.
  Interventions: Drug: Norepinephrine
- Vasopressins (Active Comparator): The vasopressin group: a group of 10 subjects that will receive vasopressin 0.04 IU/min infusion for 5 hours, starting 60 minutes before endotoxin administration.
  Interventions: Drug: Vasopressins
- Phenylephrine (Active Comparator): The phenylephrine group: a group of 10 subjects that will receive phenylephrine 0.5 μg/kg/min infusion for 5 hours, starting 60 minutes before endotoxin administration.
  Interventions: Drug: Phenylephrine
- Placebo (Placebo Comparator): The placebo group: a group of 10 subjects that will receive NaCl 0.9% infusion for 5 hours, starting 60 minutes before endotoxin administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Norepinephrine — Noradrenaline is an endogenous catecholamine with sympathomimetic effects. It has mainly α-adrenergic receptor selectivity but also β-effects in higher concentrations. It will be administered at 0.05 μg/kg/min, a clinical relevant dose on the low end of the scale.
  Other Names: Noradrenaline
  Arms: Norepinephrine
Drug: Phenylephrine — Phenylephrine is a selective α-adrenergic receptor agonist. It will be administered at 0.5 μg/kg/min, based on its relative vasopressor potency in comparison with noradrenaline.
  Arms: Phenylephrine
Drug: Vasopressins — Vasopressin is 8-arginine-vasopressin, a synthetic analogue of endogenous nonapeptide hormone. It exerts its action via V1 receptors (ubiquitous vasoconstriction) and V2 receptors (renal water resorption). It will be administered at 0.04 IU/min, a clinically relevant dose.
  Other Names: Argipressin
  Arms: Vasopressins
Drug: Placebo — NaCl 0.9% infusion
  Other Names: NaCl 0,9%
  Arms: Placebo

SUMMARY:
Noradrenaline is a catecholamine and the cornerstone treatment for the improvement of hemodynamic parameters in septic shock. Catecholamines exert profound immunomodulatory effects. Noradrenaline in vitro inhibits LPS-induced pro-inflammatory cytokine production, however, the actions on immune function in vivo have not been assessed. Furthermore, effects on the immune system of viable vasopressor alternatives for the treatment of septic patients, namely phenylephrine and vasopressin, need to be established in humans in vivo.

DETAILED DESCRIPTION:
Rationale:

Septic shock is a major medical challenge associated with a high mortality rate and increasing incidence. It has become clear that the majority of septic patients do not succumb to an initial pro-inflammatory "hit", but at a later time-point in a pronounced immunosuppressive state, so called 'immunoparalysis'. Noradrenaline is a catecholamine and the cornerstone treatment for the improvement of hemodynamic parameters in septic shock. However, catecholamines exert profound immunomodulatory effects which have mainly been studied for adrenaline. It profoundly inhibits LPS-induced production of TNF-α, and enhances production of anti-inflammatory IL-10 in vitro, as well as in animal and human models of inflammation. Although in vitro studies have shown that noradrenaline inhibits LPS-induced pro-inflammatory cytokine production as potently as adrenaline, the effects of noradrenaline on the immune system in vivo have not yet been studied. Furthermore, effects on the immune system of viable vasopressor alternatives for the treatment of septic patients, namely phenylephrine and vasopressin, need to be established in humans in vivo.

Objective: To investigate whether noradrenaline exerts immunomodulatory effects in humans in vivo and to compare noradrenaline to other vasopressors (phenylephrine and vasopressin).

Study design: A randomized double-blind placebo-controlled study in healthy human volunteers during experimental endotoxemia.

Study population: 40 healthy male volunteers, aged 18-35 yrs.

Intervention:

1. The noradrenaline group (n= 10): subjects that will receive intravenous infusion of noradrenaline 0.05 μg/kg/min for 5 hours, starting 60 minutes before intravenous administration of 2 ng/kg LPS.
2. The phenylephrine group (n=10): subjects that will receive intravenous infusion of phenylephrine 0.5 μg/kg/min for 5 hours, starting 60 minutes before intravenous administration of 2 ng/kg LPS. .
3. The vasopressin group (n = 10): subjects that will receive intravenous infusion of vasopressin 0.04 IU/min for 5 hours, starting 60 minutes before intravenous administration of 2 ng/kg LPS.
4. The placebo group (n = 10): subjects that will receive intravenous infusion of NaCl 0.9% for 5 hours, starting 60 minutes before intravenous administration of 2 ng/kg LPS.

Main parameters/endpoints:

The difference of LPS-induced TNF-α plasma concentrations following endotoxemia between the noradrenaline and the placebo groups

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥18 and ≤35 yrs
* Male
* Healthy

Exclusion Criteria:

* Use of any medication
* Smoking
* Previous spontaneous vagal collapse
* History of atrial or ventricular arrhythmia
* (Family) history of myocardial infarction or stroke under the age of 65 years
* Cardiac conduction abnormalities on the ECG consisting of a 2nd degree atrioventricular block or a complex bundle branch block
* Hypertension (defined as RR systolic > 160 or RR diastolic > 90)
* Hypotension (defined as RR systolic < 100 or RR diastolic < 50)
* Renal impairment (defined as plasma creatinin >120 μmol/l)
* Liver enzyme abnormalities
* Medical history of any disease associated with immune deficiency
* CRP > 20 mg/L, WBC > 12x109/L, or clinically significant acute illness, including infections, within 4 weeks before endotoxin administration
* Participation in a drug trial or donation of blood 3 months prior to the LPS challenge
* Use of recreational drugs within 7 days prior to experiment day
* Recent hospital admission or surgery with general anaesthesia (<3 months)
* Known anaphylaxis or hypersensitivity to the study drugs or their excipients
* Recent anaesthesia with halogenated agents
* Known cardiovascular disease (coronary artery disease)
* Known chronic nephritis

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
concentration plasma TNFalpha (pg/ml) following endotoxemia between the noradrenaline and the placebo groups | 1 day
  comparison of subjects treated with noradrenaline compared to subjects treated with placebo

SECONDARY OUTCOMES:
concentration plasma IL-6 (pg/ml) | 1 day
  Measured with Luminex assay
concentration plasma IL-8 (pg/ml) | 1 day
  Measured with Luminex assay
Leucocyte counts and differentiation | 1 day
  Measured with Luminex assay
-The phenotype of circulating leukocytes | 1 day
  Measured with Luminex assay
concentration plasma IL-10 (pg/ml) | 1 day
  Measured with Luminex assay
concentration plasma IL-1RA (pg/ml) | 1 day
  Measured with Luminex assay
concentration plasma IL-1beta (pg/ml) | 1 day
  Measured with Luminex assay
symptoms during endotoxin day | 1 day
  6 point likert scale
blood pressure | 1 day
  mmHg
temperature | 1 day
  tympanic temperature
cytokine production after ex vivo stimulation of leukocytes | 1 day
phenotype of circulating leucocytes | 1 day
Heart rate variability | 1 day
  Comparison between Holter and 2 phone applications
Breathing frequency (breaths/ min) | 1 day
  comparison between pulseoximeter and a health Patch device and VISI mobile device
Stress Levels (in percentage based on heart rate and heart rate variability) | 1 day
  Comparison between health patch device, and 2 phone applications and a subjective stress questionaire
Mean flow velocity of the median cerebral artery | 1 day
  As measured via Transcranial Doppler Ultrasound
cerebral microcirculatory flow | 1 day
  As measured via Near Infrared Spectroscopy
Tranfer function analysis | 1 day
  As derived from transcranial Doppler Ultrasound
Cerebral vascular resistance | 1 day
  As derived from transcranial Doppler Ultrasound
Cerebral Critical closing pressure | 1 day
  As derived from transcranial Doppler Ultrasound
Microvascular flow (microvascular flow index) | 1 day
  Measured via Sidestream Darkfield Imaging
Pulsatility index of the median cerebral artery | 1 day
  As measured via Transcranial Doppler Ultrasound
Mean flow index | via 1 day
  As measured via Transcranial Doppler Ultrasound
cerebral oxygenation | 1 day
  As measured via Near infrared spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Roeland Stolk, MD, Principal Investigator — Radboudumc, Intensive Care
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stolk RF, Reinema F, van der Pasch E, Schouwstra J, Bressers S, van Herwaarden AE, Gerretsen J, Schambergen R, Ruth M, van der Hoeven HG, van Leeuwen HJ, Pickkers P, Kox M. Phenylephrine impairs host defence mechanisms to infection: a combined laboratory study in mice and translational human study. Br J Anaesth. 2021 Mar;126(3):652-664. doi: 10.1016/j.bja.2020.11.040. Epub 2021 Jan 20. PMID 33483132
- [Derived] van Loon LM, Stolk RF, van der Hoeven JG, Veltink PH, Pickkers P, Lemson J, Kox M. Effect of Vasopressors on the Macro- and Microcirculation During Systemic Inflammation in Humans In Vivo. Shock. 2020 Feb;53(2):171-174. doi: 10.1097/SHK.0000000000001357. PMID 31008870